CLINICAL TRIAL: NCT01086137
Title: Assessing Salivary Biomarkers for Risk Stratification in Metabolic Syndrome
Brief Title: Biomarkers of Metabolic Syndrome and Prediabetes
Status: Completed | Type: Observational
Sponsor: West Virginia School of Osteopathic Medicine (Other)
Responsible Party: Principal Investigator, Kristie Bridges, Associate Professor, West Virginia School of Osteopathic Medicine
Other Study IDs: BCS-100.1; KB01082010 (Other: WVSOM)
Record Dates: First submitted 2010-03-11; First posted 2010-03-12 (Estimated); Last update posted 2013-08-07 (Estimated); Status verified 2013-08

CONDITIONS: Metabolic Syndrome; Diabetes; Prediabetes; Hypertension
Keywords: salivary biomarker; metabolic syndrome; prediabetes; diabetes hypertension
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus; Prediabetic State; Hypertension

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — saliva

SUMMARY:
The purpose of this study is to investigate the feasibility of using salivary biomarkers to screen for complications of metabolic syndrome including prediabetes.

ELIGIBILITY:
Inclusion Criteria:

* Between the ages of 18 and 65 years
* Males and females will be included in this study
* All ethnic backgrounds will be included in this study
* Acceptable health based on interview and medical history
* Ability to comply with requirements of the study
* Ability and willingness to provide signed informed consent

Exclusion Criteria:

* Eating or drinking anything but water within 10 hours of sample collection
* Autoimmune disease
* Type 1 diabetes
* Pregnancy (< 6 weeks postpartum)
* History of Sjorgren's Syndrome
* Dental work within the last two weeks
* Ongoing or active parasitic, fungal, viral or bacterial infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: community sample
Sampling Method: Non-Probability Sample
Enrollment: 102 (Actual)
Dates: Start 2010-03; Primary Completion 2011-12 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
Salivary Biomarker Levels | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Kristie G Bridges, PhD, Principal Investigator — WVSOM
Locations (1):
- West Virginia School of Osteopathic Medicine, Lewisburg, West Virginia, United States